CLINICAL TRIAL: NCT06978439
Title: Rivaroxaban in Chinese Children With Giant Coronary Artery Aneurysm After Kawasaki Disease: a Pilot Study
Brief Title: Model-informed Dose Optimization for Rivaroxaban in Children With Giant Coronary Artery Aneurysm After Kawasaki Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIVA-KD-pilot
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Kawasaki Disease; Pilot Study; Coronary Artery Aneurysm; Rivaroxaban
Keywords: kawasaki disease; giant coronary artery aneurysm; rivaroxaban; model-informed dose optimization; anticoagulant
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rivaroxaban (Experimental): Rivaroxaban as anticoagulant will be administered for children with giant coronary artery aneurysm after Kawasaki disease. The initial dosing regimen of rivaroxaban is a 15 mg-equivalent, age and bodyweight-adjusted dosing regimen, which was proposed by the model-informed dose optimization study.
  Interventions: Drug: Rivaroxaban (Xarelto)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto) — Administered in an age- and bodyweight-adjusted, 15 mg-equivalent dose regimen proposed by model-informed dose optimization study
  Other Names: Anticoagulation

SUMMARY:
Based on a population pharmacokinetic model-based dose optimization study, a 15 mg-equivalent, age-, and bodyweight-adjusted dosing regimen for Chinese children with giant coronary artery aneurysms after Kawasaki disease was proposed. This single-center, single-arm, pilot study aims to evaluate the feasibility of the 15 mg-equivalent dosing regimen within a limited sample size.

Patients will be followed for more than 6 months. Clinical outcomes, including coronary artery thrombosis, major adverse cardiovascular events, and bleeding events, will be recorded. Rivaroxaban levels will be measured to assess the robustness of the model-informed dose optimization.

DETAILED DESCRIPTION:
Giant coronary artery aneurysm (GCAA) is a rare but severe cardiac complication of Kawasaki disease (KD). Due to the abnormal blood rheology and the hyper-inflammatory response accompanied by thrombocytosis during the acute phase, patients with GCAA are at high risk of coronary artery thrombosis and major adverse cardiovascular events.In such instances, lifelong antiplatelet (aspirin or clopidogrel) and anticoagulant therapy (warfarin or low molecular weight heparin, LMWH) may become necessary.

In 2022, two compounds, the direct activated Factor X (FXa) inhibitor rivaroxaban was approved by international regulatory agencies for two specific pediatric indications, supported by pharmacometrics models. For instance, a dosing regimen matching exposures of 20 mg daily in adults (the 20 mg-equivalent dosing regimen) is indicated for children under 18 years with venous thromboembolism (VTE). Secondly, a dosing regimen matching exposures of 10 mg daily in adults (the 10 mg-equivalent dosing regimen) is indicated for post-Fontan patients aged two years or older, as shown in the UNIVERSE study, which compared rivaroxaban to aspirin. However, no trials have yet compared rivaroxaban with warfarin/LMWH in pediatric patients with GCAA after KD.

Inter-ethnic population pharmacokinetic (PPK) analyses have suggested that Asian patients may require a lower dosage of rivaroxaban, consistent with the findings from the J-ROCKET trail in Japanese adults. Accordingly, the maximum dosage for Japanese children with VTE (≥ 50 kg) has reduced from 20 mg q24h (every 24 hours) to 15 mg q24h. However, reports on rivaroxaban use in pediatric patients with GCAA after KD, especially in those from Asian countries, remains limited. Its application is more challenging due to (i) increased bleeding risk from concomitant antiplatelet drug use; (ii) the predominance of younger patients (typically < 3 years) with variability in hepatic and renal function, as well as growth and development.3 Given the low incidence of GCAA, quantitative pharmacometrics is a highly promising approach for precision dosing of rivaroxaban in these patients.

Therefore, the investigators retrospectively collected the clinical experience of rivaroxaban off-label use in Chinese pediatric patients with GCAA after KD from 2023.1 to 2023.12. With clinical evidence and model-extrapolation, the investigators conducted a quantitative pharmacometrics model-based dose optimization study and proposed a 15 mg-equivalent dosing regimen for thromboprophylaxis in Chinese children with GCAA after KD, those who require dual antithrombotic therapy.

This pilot study aims to assess the potential of rivaroxaban for thromboprophylaxis in pediatric patients with KD after GCAA. Specifically, this study seeks to: (ⅰ) preliminarily evaluate the feasibility, efficacy and safety of the 15 mg-equivalent dosing regimen in target population, (ii) provide pharmacokinetic (PK)/pharmacodynamic (PD) data on rivaroxaban in Chinese children.

ELIGIBILITY:
Inclusion Criteria:

1. Giant coronary artery aneurysm(s) in any coronary artery after acute stage of Kawasaki disease. Giant coronary artery aneurysm(s) should be confirmed by two-dimensional echocardiography and meet the diagnostic criteria of Z-score ≥10 or coronary artery internal diameter ≥8mm;
2. Anticoagulant with antiplatelet drug therapy for anti-thromboprophylaxis is recommended for the next 6 months;
3. Participant should be able to tolerate oral feeding, nasogastric or gastric feeding;
4. Children aged 1 Month to<18 years, bodyweight ≥ 2600g.

Exclusion Criteria:

1. Active bleeding or bleeding risk contraindicating anticoagulant therapy
2. With history of venous thromboembolism or risk factors related with venous thromboembolism, like congenital heart disease, carcinoma, central venous catheter or long-term immobilization.
3. Hypersensitivity or any other contraindications listed in the local labeling for the comparator treatment or experimental treatment
4. An eGFR <30 mL/min/1.73 m2 (For children younger than 1 year, serum creatinine results above 97.5th percentile)
5. Platelet count < 100 x 109/L
6. Hepatic disease which is associated with either: coagulopathy leading to a clinically relevant bleeding risk, or alanine aminotransferase > 5x ULN or total bilirubin > 2x ULN with direct bilirubin > 20% of the total
7. Sustained uncontrolled hypertension defined as systolic and/or diastolic blood pressure >95 th age percentile
8. Concomitant use of strong inhibitors of both CYP3A4 and P-glycoprotein, including but not limited to all human immunodeficiency virus protease inhibitors and the following azole-antimycotics agents: ketoconazole, itraconazole, voriconazole, posaconazole, if used systemically (fluconazole is allowed)
9. Concomitant use of strong inducers of CYP3A4, including but not limited to rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine
10. Hypersensitivity or any other contraindications listed in the local labeling for the comparator treatment or experimental treatment
11. Inability to cooperate with the study procedures and follow-up visits
12. Refuse to provide informed consent

eGFR, estimated glomerular filtration rate; ULN, upper level of normal; TB, total bilirubin (TB); CYP3A4, cytochrome P450 isoenzyme 3A4

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of new thrombosis in coronary arteries | From enrollment to the 6th month after treatment
  It is a binary variable. Every echocardiography conducted during study period will be assessed and documented. Investigators will evaluate whether new thrombosis occurs in coronary arteries.
Composite of Major bleeding or Clinically relevant non-major bleeding event | From enrollment to the 6th month after treatment
  It is a binary variable. Major bleeding is defined as 1.Fatal bleeding; 2.Clinically overt bleeding associated with a decrease in Hgb of ≥20 g/L (2 g/dL) in a 24-h period; 3.Critical site bleeding, such as retroperitoneal, pulmonary, pericardial, intracranial, or otherwise involves the central nervous system; 4.Bleeding that requires an intervention via an invasive procedure; 5.Overt bleeding for which a reversal agent is administered. Clinically relevant non-major bleeding event is defined as 1.Bleeding that results in a medical or procedural intervention not meeting major bleeding criteria, including a medication change (reducing, holding, or changing anticoagulation or addition of new medication) ; 2.Bleeding that results in hospitalization or increased level of care; 3.Overt bleeding for which a blood product is administered, and does not meet the criteria for major bleeding

SECONDARY OUTCOMES:
Occurrence of major adverse cardiovascular event | From enrollment to the 6th month after treatment
  It is a binary variable. Major adverse cardiovascular event (MACE) includes unstable angina, acute myocardial infarction, stroke, hospitalization for heart failure, unplanned revascularization, cardiovascular death. If any of the MACEs occur during the study period, it will be recorded as 1; otherwise, it will be recorded as 0. The definition of each MACE refers to the following guidelines and consensus: 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials, 2019 European Society of Cardiology Guidelines for the diagnosis and management of chronic coronary syndromes, Fourth universal definition of myocardial infarction, and 2023 European Society of Cardiology Guidelines for the management of acute coronary syndromes.
Any adverse events | From enrollment to the 6th month after treatment
  It is a text variable. If any adverse events( including durg allergy, severe infection, hepatic dysfunction, renal dysfunction, hypertension, fatigue, abdominal pain or others) occur will be reported to the data and safety monitoring board. The detail of adverse event will be recorded, including classification of adverse event, time of occurrence, symptoms, treatment, resolution time, and outcome.
Any dose adjustments for rivaroxaban | From enrollment to the 6th month after treatment
  It is a text variable. Any dose adjustments for rivaroxaban will be recorded, including time of dose adjustment, reason for dose adjustment, dosage, and outcome. Rivaroxaban plasma concentration and rivaroxaban-calibrated anti-factor Xa activity will be measured after at least 3 consecutive doses

OTHER OUTCOMES:
Plasma concentration of rivaroxaban at specific timepoint | From enrollment to the 6th month after treatment
  Rivaroxaban plasma concentration will be measured by high performance liquid chromatography tandem mass spectrometer at specific timepoint. It includes 1. 20 minutes to 1 hour after the first dose; 2. 7 ± 1 hours after the first dose; 3. Ctrough: before the scheduled dose after at least three consecutive doses; 4. Cmax: 3 ± 1 hours after at least three consecutive doses. And Ctrough and Cmax will be re-measured after each dose adjustment.
Rivaroxaban-calibrated anti-factor Xa activity at specific timepoint | From enrollment to the 6th month after treatment
  Rivaroxaban-calibrated anti-factor Xa activity will be measured at specific timepoint. It includes 1. 20 minutes to 1 hour after the first dose; 2. 7 ± 1 hours after the first dose; 3. Ctrough: before the scheduled dose after at least three consecutive doses; 4. Cmax: 3 ± 1 hours after at least three consecutive doses. And Ctrough and Cmax will be re-measured after each dose adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Liu, MD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No